CLINICAL TRIAL: NCT04570904
Title: Broadening Our Understanding of Early Versus Late Influenza Vaccine
Brief Title: Broadening Our Understanding of Early Versus Late Influenza Vaccine Effectiveness
Acronym: BELIEVE
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); World Health Organization (Other); University of Warwick (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0787; IRAS (Other: 284733); Sponsor Reference Number (Other: UOL0787)
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2020-09

CONDITIONS: Influenza; Influenza -Like Illness
Keywords: Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — With participant consent, any unused serum samples will be stored for future ethically approved research and shared with other research collaborators in other academic institutions and industry partners inside and outside of the UK for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early HCWs: Health Care Workers vaccinated early prior to the influenza season
  Interventions: Biological: Influenza vaccination at different time points
- Late HCWs: Health Care Workers vaccinated just prior to the influenza season
  Interventions: Biological: Influenza vaccination at different time points
- Inpatients: Inpatients recruited for evaluation of new approaches to influenza diagnosis

INTERVENTIONS:
Biological: Influenza vaccination at different time points — All HCWs will receive the seasonal influenza vaccine but at two different time points.
  Groups: Early HCWs; Late HCWs

SUMMARY:
This study uses a prospective cohort design to investigate if the seasonal influenza vaccine is equally effective when given early and late before the proceeding influenza season. All health care workers will be vaccinated for seasonal influenza either 3 months before or 1 month prior to the start of the influenza season. HCWs that consent to take part in the study will have 4 blood samples taken for an antibody check. The initial antibody checks will be done just prior to vaccination as well as 2 weeks after vaccination. Subsequent samples will be taken at the peak of influenza season and at the end of the influenza season.

HCWs that develop ILI during the course of the influenza season will be asked to complete a questionnaire and oropharyngeal self-swab. HCWs will also provide exhaled breath samples and wear a mask in order to evaluate novel non-invasive methods for diagnosis of influenza.

Influenza positive and negative inpatients identified through the University of Leicester's laboratory system will also be asked to provide breath samples to evaluate this technique for the diagnosis of influenza.

DETAILED DESCRIPTION:
Recruitment, Screening and Eligibility Assessment

Potential participants (University Hospitals of Leicester NHS Trust, UHL staff) will be contacted by email to advertise and explain the study. The email will be part of the routine seasonal influenza vaccination emails which are sent out each year to remind UHL staff to be immunised. In addition, the investigators will advertise by posters in the high staff traffic areas, e.g. the restaurant, and our Occupational Health Team will assist with this advertising of the study. The investigators expect some Health care workers (HCWs) to become aware of the study through word of mouth.

The study will have two phases of recruitment. For the month of September for the 'early' vaccination group, and from mid-November to mid-December for the 'late' vaccination group - the exact timings may vary depending on when the inactivated influenza vaccines are received and the seasonality of the virus, as all recruitment will be completed prior to the start of the influenza season. Allocation to the two vaccination groups will not be randomised; it will be the HCWs decision if they would like to have the vaccination either early or late. There will be a limit of 200 HCWs recruited to each group.

Individuals who express an interest in taking part in the study will be given an information sheet either in person or via email. Following this the investigators will give them as long as they need to decide whether or not to participate in the study. If the individual agrees to participate, a member of the research team will screen and confirm eligibility. Participants will only be recruited if all criteria are satisfied. At this time arrangements will be made for staff members to attend an initial appointment at the Research Space at the LRI. Recruitment in the research area will comply with the current social distancing measures in place at UHL.

At this initial appointment the study will be explained to staff members in groups. A member of the research team will then seek written informed consent as detailed below from each HCW individually. If an individual has more questions about the study another study team member will be allowed to support and facilitate informed consent.

Recruitment of inpatients Clinicians on the acute medical wards will be notified prior to the start of the influenza season via email and posters, in clinical areas, of the study involving inpatients with (influenza like illness) ILI. University Hospitals of Leicester Virology department routinely call the clinical team of positive influenza cases in inpatients during the influenza season. When the clinical team then goes to explain this diagnosis to the patient they would also make them aware of the study and provide them with a participant information leaflet. Following this the investigators will give the patient as long as they need to decide whether or not to participate in the study. If the individual agrees to participate they will inform a member of the clinical team who will then notify the research team. A member of the research team will attend the ward to screen and confirm eligibility. Participants will only be recruited if all criteria are satisfied. Using laboratory results data, twenty inpatients with confirmed influenza-negative swabs will also be recruited in the same way, as a control group.

Study Visits

The following activities will be carried out at each visit and recorded in the CRF:

Visit 1: Baseline visit

* Participants will be enrolled providing they meet inclusion and exclusion criteria and give fully informed, written consent.
* Participants will then be assigned a study number
* Participants will complete a short questionnaire which will include demographic information: Age, sex, ethnicity, job role, medical co-morbidities, regular medications, smoking history, history of influenza infections and influenza vaccine.
* Collect 10ml clotted blood pre-immunisation for baseline antibodies. Process blood and store serum for serology assays. The influenza vaccine will be administered in the normal way.
* Participants will be given a thermometer, two influenza self-sampling kits (i.e. a swab and a viral transport medium tube with a Microbiology sample bag), and two information forms that they will complete in the event that they develop any influenza-like illness (ILI). An ILI will be defined as per the WHO case definition as a fever of >37.8oC and cough with onset within the last 10 days. They will be shown how to operate the thermometer, take a self-swab (i.e. a throat swab), and how to secure the swab in the sampling tube. They will also be show how to complete an ILI event form (ILIef) - briefly recording the timing and nature of their ILI symptoms/signs.

Visit 2: 3 weeks after baseline visit (+ or - 7days)

* Collect 10ml clotted blood for serology. Process blood and store serum.
* Participants will be asked to provide breath samples, this will act as a control against which breath samples that occurred during ILI will be compared Visit 3: Peak influenza season usually January to February (+ or - 30 days)
* Collect 10ml clotted blood for serology. Process blood and store serum. Visit 4: End of influenza Season usually April to May (+ or - 30 days)
* Collect 10ml clotted blood for serology. Process blood and store serum. ILI event study visit Study participants will contact the study team by email or phone to alert them that an ILI event has occurred, and to arrange for a study team member to collect the swab and ILIef from them, as soon as possible after it has been taken, for appropriate storage (in a -80oC freezer) until tested. If study participants are at home when they develop ILI they will be asked to complete the self-swab and ILef. The swab will be doubled bagged and collected by a member of the research team in accordance with the transport guidance issued in the Government's guidance on COVID-19: safe handling and processing for samples in laboratories in accordance with UN3373, packing instructions 650. Swabs will be delivered to the UHL virology laboratory and processed according to standard operating procedures (see Section 8.7.1).

It will be reiterated to the study participant that results of these swab results will be emailed and phoned through to them along with the latest occupational health advice. They will be advised to follow occupational health policy for ILI whilst awaiting the swab results, report sickness in the normal way and contact their GP if further medical advice regarding this current period of illness is needed.

The contents of the ILIef will be entered into the participants case report form (CRF), no personal information will be included. These details will be used in the interpretation of the viral sequencing and antibody titres, performed at WHO Melbourne.

If the study participant is at work when they develop ILI they will be asked to provide a breath sample and mask sample for the detection of influenza using novel methods prior to leaving work. Sampling materials will be brought to where the HCW is located but if this could not happen straight away then the HCW would be told to follow occupational health advice and go home. Specimens collected from these processes are detailed in section 8.7.

Inpatient breath sample Inpatients will be approached as per the usual UHL infection control policy. Only patients who have results available for a recent throat swab tested for common respiratory pathogens will be approached. COVID-19 positive wards will not be involved in recruitment instead inpatients with Influenza and other respiratory viruses will be recruited from COVID-19 negative wards. Patients who are confirmed influenza positive are usually managed in side rooms as per policy. In all cases, the patient will not be required to come into contact with the analysis equipment, as the breath capture and analytical processes are separate. Mask sampling will not be undertaken on patients who require oxygen therapy via a face mask. Once consented to the study one member of the research team will approach the patient with the masks, syringes and mouthpieces needed for breath sample collection. A repeat throat swab will also be taken at this time so accurate comparison can take place between the novel diagnostic methods and current practise. All three breath sampling methods, where possible, will be used. Once the samples have been collected they will be placed in a biological hazard bag and taken to the analysis machines. Swabs and mask samples will be transported to the virology Laboratory at Leicester Royal Infirmary for processing. The breath capture equipment (syringes and disposable mouth pieces) will be disposed of in the normal way for clinical waste. TD tubes and the Bio-VOC sampler will be double bagged and will be decontaminated. This is the only study visit required by inpatients and no further follow up is required.

Self-swabs The swabs will be delivered to the Department of Clinical Microbiology at University Hospitals of Leicester NHS Trust where they will be handled under Cat 2 (BSL-2) conditions. They will be vortexed, and swabs discarded leaving the inoculated virus transport medium (VTM). The VTM tubes will be tested on a standard diagnostic assay (routinely used for hospital patient testing) to check for the presence of influenza (as many different respiratory viruses can cause an 'influenza-like illness'). If influenza is detected, then an aliquot of this VTM will be sent to WHO Melbourne, along with the serum samples, for viral sequencing of influenza. VTM will be transported to the WHO laboratory under UN3733/Category B regulations.

VOC breath analysis All three analysis platforms will use the same basic collection approach. Participants will be asked to not to have eaten or drank anything at least 30 minutes before breath sampling. Prior to sampling swill their mouth with water which they can then swallow - and then provide three non-forced breath samples by exhaling into disposable mouthpieces for 3-5 seconds. Researchers will wear PPE dictated by local trust policy at UHL for collecting nasal and oral swabs. Disposable clinical gloves will be used for all procedures. The analytical devices will be kept on the ward or in a research area away from direct patient contact.

For GC-IMS analysis, the mouthpiece is attached to a 10cm long plastic tube. As the patient exhales into the tube, the researcher will draw a breath sample into a 5ml syringe part way down the tube.

The sample will then be injected from the syringe by the researcher into the BreathSpecTM GC-IMS device for analysis. Any infectious material contained within the sample will be destroyed by being heated to over 60°C as part of the analytical process.

The eNose uses a commercial CE marked breath capture unit, the Markes Bio-VOC. The unit holds 129ml of breath, comes sealed and only opened when ready to use, and is disposable. The user fits a cardboard mouthpiece to the unit prior to sampling. Once the patient has breathed into the unit the mouthpiece is removed and a syringe fitting is added, which connects to the eNose. The syringe is then depressed and the sample is analysed. Analysis time is under 5 minutes. The eNose machine will be decontaminated at the end of each day of use according to the manufacture's guidelines.

For GC-MS analysis, a further breath sample is again collected using the Markes Bio-VOC unit as above. Once the sample is collected it will be transferred onto a thermal desorption (TD) tube (typically 89mm x 6.4mm). The inner walls of the tube are coated with an absorbent layer to which breath chemicals adhere. The TD tube is placed at the end of the Bio-VOC unit and captured air is pushed through the tube. Once completed, the ends of the tubes are sealed with end caps. A validated decontamination process is then undertaken for the Bio-VOC sampler and TD tubes through a long / high heat cycle to ensure the virus is killed off. The decontaminated TD tubes will be kept in storage boxes in the research area of Leicester Royal Infirmary for transport to the University of Warwick for analysis and final disposal, as per a pre-defined Material Transfer Agreement.

The results of the GC-IMS analysis will be uploaded regularly from the BreathSpecTM onto a DataSync shared drive and downloaded by analysts at the University of Warwick. No identifiable data will be associated with this data, only a study number.

Mask sampling Mask sampling consists of participants wearing a modified face mask (flat surgical, duckbilled or FFP1) which contains up to 5 strips of 3D printed Polyvinyl alcohol (PVA) for up to 60 minutes whilst being observed by a member of the research team. The investigators will provide training, support and personal protective equipment to research staff obtaining samples and agree protocols for local processing. Prior to use masks are sterilised and kept in sealed sample bags, once worn they are placed back in these bags and sealed. They will be transported to the UHL Virology Laboratory in line with current Risk Assessments and Standard Operating procedures concerning transporting hazardous materials. Viral RNA will be extracted and quantified from the PVA strips within the masks using Real-Time quantitative PCR. The processing of the PVA strips requires them to be dissolved into water, from which the RNA virus is extracted and analysed using molecular methods. The masks and bags will be destroyed.

Serum testing and viral sequencing On each of the scheduled days requiring serum samples, the clotted blood will be stored at 2oC to 8oC and centrifuged within 24 hours at the Research Space, LRI. Sera will be stored in cryovials, with all cryovials labelled with the participant's study number, visit number and date of collection at the Research Space, LRI. Samples will be stored frozen at -80 oC until shipment. One set of cryovials will be sent to the WHO reference laboratory in Melbourne once all samples have been collected. The other set of cryovials will be stored as a safety measure in case of transport issues. With participant consent, any unused serum samples will be stored for future ethically approved research and shared with other research collaborators in other academic institutions and industry partners inside and outside of the UK for future research. Serum will be used for Hemagglutination inhibition and microneutralization assays and once all samples have been processed results will be sent back to the research team at Leicester.

Haemagglutination Inhibition (HAI) and Microneutralisation (MN) assays, together with influenza viral sequencing will be performed at the WHO Collaborating Centre for Reference and Research on Influenza (VIDRL), Peter Doherty Institute for Infection and Immunity, 792 Elizabeth Street, Melbourne, VIC 3000, Australia.

ELIGIBILITY:
Inclusion Criteria:

For Health care workers (HCWs)

* Willing and able to give informed consent
* Employee at the University Hospitals of Leicester
* Willing and able to have the inactivated Influenza vaccine
* Age ≥16 For inpatients
* Inpatient at University Hospitals of Leicester
* Throat swab for influenza completed in the last 72 hours
* Willing and able to give informed consent
* Well enough to provide an exhaled breath sample without causing distress or discomfort
* Well enough to wear a face mask without causing distress or discomfort
* Age ≥16

Exclusion Criteria:

* Age <16
* Unwilling and/or unable to give informed written consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be composed of HCWs at University Hospitals of Leicester, that are eligible for the seasonal influenza vaccine A further study population will be composed of inpatients at the University Hospitals of Leicester presenting and / or admitted with Influenza like illness
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Difference in antibody titre | Antibody titres to be analysed at the end of the study once all samples collected - estimated May 2021
  Difference in antibody titres at set time points during the 2020/21 influenza season in HCWs stratified by those who are vaccinated early and late

SECONDARY OUTCOMES:
Influenza infections | Influenza positive swabs to be analysed at the end of the study once all samples collected - estimated May 2021
  The number of laboratory-confirmed influenza infections by real time PCR in HCWs vaccinated early and late
Breath analysis for influenza diagnosis | Results to be analysed post influenza season - estimated May 2021
  The detection of markers of influenza infection in breath samples using GC-IMS, eNose and GC-MS
Mask sampling for influenza diagnosis | Results to be analysed post influenza season - estimated May 2021
  The detection of influenza by PCR using a novel mask sampling technique

CONTACTS AND LOCATIONS:
Overall Officials: Manish Pareek, PhD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Royal Infirmary, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The participants will be identified only by initials and a participant ID number on the CRF and any electronic database. All documents will be stored securely and only accessible by study staff and authorised personnel. The study will comply with the Data Protection Act which requires data to be anonymised as soon as it is practical to do so.

REFERENCES:
- [Derived] Nazareth J, Barr I, Sullivan SG, Goss C, Pan D, Martin CA, Sahota A, Stephenson I, Tang JW, Pareek M. Intra-season waning of immunity following the seasonal influenza vaccine in early and late vaccine recipients. J Infect. 2022 Dec;85(6):e172-e174. doi: 10.1016/j.jinf.2022.10.011. Epub 2022 Oct 13. No abstract available. PMID 36243199